CLINICAL TRIAL: NCT00002508
Title: INTENSIVE CHEMOTHERAPY FOR RELAPSED OR REFRACTORY GERM CELL TUMORS EMPLOYING HIGH-DOSE CARBOPLATIN, ETOPOSIDE, AND THIOTEPA WITH AUTOLOGOUS BONE MARROW RESCUE FOR PATIENTS 15 TO 60 YEARS OF AGE
Brief Title: Combination Chemotherapy Followed by Bone Marrow or Stem Cell Transplantation in Treating Patients With Relapsed or Refractory Germ Cell Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: Fox Chase Cancer Center (Other)
Responsible Party: Temple University Bone Marrow Transplant Program, Temple University health Systems
Purpose: Treatment
Other Study IDs: CDR0000078063; TUHSC-1839; NCI-V92-0204
Record Dates: First submitted 1999-11-01; First posted 2004-03-11 (Estimated); Last update posted 2010-10-01 (Estimated); Status verified 2010-09

CONDITIONS: Extragonadal Germ Cell Tumor; Ovarian Cancer; Testicular Germ Cell Tumor
Keywords: recurrent malignant testicular germ cell tumor; recurrent ovarian germ cell tumor; extragonadal germ cell tumor
MeSH Terms: conditions — Ovarian Neoplasms; Testicular Germ Cell Tumor; Testicular Neoplasms | interventions — Carboplatin; Etoposide; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Drug: carboplatin
Drug: etoposide
Procedure: autologous bone marrow transplantation
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Peripheral stem cell transplantation may allow doctors to give higher doses of chemotherapy and kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of combination chemotherapy followed by peripheral stem cell transplantation or bone marrow transplantation in treating patients who have relapsed or recurrent germ cell cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate, overall survival, and disease-free survival of patients with refractory or relapsed germ cell carcinoma treated with high-dose induction chemotherapy comprising carboplatin and etoposide followed by autologous bone marrow or peripheral blood stem cell rescue.

OUTLINE: Autologous peripheral blood stem cells (PBSC) or bone marrow is harvested. Patients receive carboplatin IV continuously and etoposide IV over 1 hour on days -5 through -3. Autologous PBSC or bone marrow is reinfused on day 0.

PROJECTED ACCRUAL: A maximum of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Documented relapsed or refractory germ cell cancer of the following sites of origin: Testes Ovary Retroperitoneum Mediastinum Other sites Any stage of disease allowed Any histologic subtype allowed Seminoma only allowed if ineligible for radiotherapy Failed to achieve complete remission (CR) following at least 3 courses of a standard platinum-containing regimen or experienced clear relapse following CR obtained with such a regimen Absence of tumor markers in the presence of stable residual masses after initial treatment may be allowed (surgical biopsy should be performed; if medically safe, to confirm persistence of disease and rule out mature teratoma or fibrosis) Prior CNS involvement allowed in the absence of gross residual CNS tumor following definitive local therapy (surgery plus radiotherapy) No gross tumor involvement on bone marrow biopsy

PATIENT CHARACTERISTICS: Age: 15 to 60 Performance status: Karnofsky 80-100% Hematopoietic: Granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 2.0 mg/dL SGOT/SGPT less than 2 times normal Albumin greater than 3.0 mg/dL Renal: Creatinine less than 1.8 mg/dL Cardiovascular: LVEF at least 50% No other serious cardiac disease that would preclude transplantation Pulmonary: DLCO, FEV1, and FVC at least 50% predicted pO2 at least 70 mm Hg on room air Other: HIV negative No other concurrent serious psychiatric, neurologic, neoplastic, immunologic, or other medical problem that would preclude transplantation Not pregnant

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics No prior chest irradiation Surgery: See Disease Characteristics

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 1990-11; Primary Completion 2001-09 (Actual); Study Completion 2001-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R. Klumpp, MD, Study Chair — Fox Chase Cancer Center
Locations (1):
- Temple University Cancer Center, Philadelphia, Pennsylvania, United States